CLINICAL TRIAL: NCT02662127
Title: Local Endogenous Biomarkers in the Later Stages of Chronic Venous Disease Versus Controls During Gravitational Stress, Prolonged Elevation Recovery and Compression
Brief Title: Effect of Standing, Lying and Stockings on Blood Bio-markers (v.1)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: London North West Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 198127
Record Dates: First submitted 2016-01-13; First posted 2016-01-25 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: Chronic Venous Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SIGVARIS®. Class 2 - RAL: 23-32 (Experimental): Graduated elastic compression stockings
  Interventions: Device: SIGVARIS® Class 2 - RAL: 23-32.

INTERVENTIONS:
Device: SIGVARIS® Class 2 - RAL: 23-32. — Below knee graduated elastic compression stocking

SUMMARY:
Venous disease effects 25% of the population and most healthy people experience venous symptoms after standing for too long. The prime function of leg veins is drainage. Failure leads to a condition called chronic venous insufficiency (CVI) with leg pain, heaviness, swelling, varicose veins, ankle skin changes, eczema and occasionally venous ulcers. The aim of the study is to identify blood components (biomarkers) that occur during the damaging phase of standing versus the healing phases of lying recovery and with medical compression stockings. This will be achieved by taking a blood sample from the ankle region at 3 separate visits (days) to the vascular laboratory at Ealing Hospital. The first visit will be after supervised standing for 1 hour. The second after supervised lying and the third standing whilst wearing a medical compression stocking. Healthy volunteers will be compared to patients with advanced CVI.

The potential importance to patients and the public is threefold. Firstly, biomarker profiles will be obtained in each of the 3 states to increase understanding in the cellular mechanisms of damage and recovery. In this way "bad" and "good" biomarkers can be identified. Secondly, drug treatments may develop from this research to adjust biomarkers towards a favourable profile. Thirdly, the success of treating CVI with surgery, venous intervention or compression can be monitored. Whilst it is known that relief of gravitational stress is the treatment for all forms of CVI, the mechanisms of repair and its discrimination from damage have yet to be identified.

DETAILED DESCRIPTION:
It is well known that graduated elastic compression stockings (GECs) provide a favourable environment by off-setting the damaging effects of dependency, reducing leg oedema, preventing leg ulceration and in symptom relief. On a haemodynamic level, their mechanism of action in augmenting the venous return has been quantified. However, on a molecular level, their action in modulating local endogenous biomarkers towards a favourable profile is poorly understood. This requires further investigation.

Our hypothesis is that there are two types of biomarkers: (i) damaging inflammatory biomarkers which are increased after prolonged gravitational dependency, (i) healing reparative biomarkers which are increased after prolonged elevation recovery. Local venous blood samples draining the area of investigation may be more representative of loco-regional processes than systemic blood samples from the arm.

This is a single centre, collaborative, interventional, controlled, proof-of-concept trial.

The primary aim of this study is to investigate the effect of GEC stockings on modulating biomarkers towards a healing profile.

Planned interventions:

There will be 4 study visits per subject.

1. Recruitment, patient selection, distribution of information leaflets and consent form, explanation of the demands of the study, claiming of expenses, duplex scanning and visit scheduling.
2. Formal consent. Blood test. The stage of "damage" will be in the afternoon after standing all morning plus an hour of extra standing in the laboratory.
3. Blood test. The stage of "healing" will be in the morning after nocturnal sleep plus an hour of extra elevation (20 degrees elevated from supine) in the laboratory.
4. Blood test. The stage of "treatment" will be from the effects of a class II below knee stocking after standing all morning plus an hour of extra standing in the laboratory.

All venous blood will be taken from the ankle region. The samples will be taken during a gravitational stress, after elevation recovery and after the therapeutic effect of the compression stocking. These specifications must be met with due care and diligence to ensure that the results are meaningful. The samples will be collected in citrated tubes, centrifuged at 5,000 rpm for 10 minutes to achieve platelet poor plasma and stored at -20 degrees for batch analysis.

Proposed biomarkers for quantification:

Radox (IL-2, IL-4, IL-6, IL-8, IL-10, VEGF, IFNγ, TNFα, IL-1α, IL-1β, MCP-1, EGF) and D-dimer.

Matrix metalloproteinases (MMP-1, MMP-2, MMP-3, MMP-7, MMP-8, MMP-9, MMP-10, MMP-12 and MMP-13) and also 4 tissue inhibitors of MMPs (TIMP-1, TIMP-2, TIMP-3 and TIMP-4).

ELIGIBILITY:
Inclusion Criteria:

1. Patients from the vascular clinic at Ealing Hospital with venous disease

   1. Venous skin changes including lipodermatosclerosis and pigmentation
   2. Significant reflux >0.5 seconds on duplex
2. Volunteers from NHS healthcare workers or the general public

   1. Absence of venous symptoms
   2. Freedom from varicose veins or skin changes

Exclusion Criteria:

1. Previous treatment for varicose veins on the study leg
2. Previous history of deep or superficial vein thrombosis
3. Receiving anticoagulation
4. Haematological disorders of coagulation or thrombosis
5. Pregnancy
6. Significant peripheral vascular disease
7. Cardiac failure or orthopnoea
8. Uncontrolled/active malignancy
9. Significant impairment of mobility
10. Connective tissue or autoimmune disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Number of biomarkers which decrease greater than 20% of the baseline level as a result of the interventions of (i) lying down and with a (ii) stocking | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Evi Kalodiki, MD PhD FRCS, Principal Investigator — London North West Healthcare NHS Trust
Locations (1):
- Ealing Hospital, LNWH NHS Trust, Ealing, United Kingdom

IPD SHARING:
Plan to Share IPD: No